CLINICAL TRIAL: NCT01353430
Title: Characterization of Familial Myopathy and Paget Disease of Bone
Brief Title: Characterization of Inclusion Body Myopathy Associated With Paget's Disease of Bone and Frontotemporal Dementia (IBMPFD)
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Virginia Kimonis, Professor, University of California, Irvine
Other Study IDs: #20075832
Record Dates: First submitted 2011-01-26; First posted 2011-05-13 (Estimated); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Inclusion Body Myopathy With Early-onset Paget Disease and Frontotemporal Dementia; Paget Disease of Bone; Frontotemporal Dementia; Myopathy
Keywords: IBMPFD - Inclusion Body Myopathy associated with; Paget's disease of bone and Frontotemporal Dementia; VCP gene - Valosin-containing protein gene
MeSH Terms: conditions — Inclusion Body Myopathy With Early-Onset Paget Disease And Frontotemporal Dementia; Osteitis Deformans; Frontotemporal Dementia; Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, skin and muscle biopsy, urine sample, if available samples obtained from previous diagnostic evaluations such as muscle biopsy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VCP families: Patients with a personal or family history of VCP associated disease.

SUMMARY:
The investigators are researching families with inherited inclusion body myopathy (IBM) and/or Paget disease of bone (PDB) and/or dementia (FTD) which is also called IBMPFD. IBMPFD is caused by mutations in the VCP gene. Our main goal is to understand how changes in the VCP gene cause the muscle, bone and cognitive problems associated with the disease.

The investigators are collecting biological specimen such as blood and urine samples, family and medical histories, questionnaire data of patients with a personal or family history of VCP associated disease. Participants do not need to have all symptoms listed above in order to qualify. A select group of participants may be invited to travel to University of California, Irvine for a two day program of local procedures such as an MRI and bone scan.

Samples are coded to maintain confidentiality. Travel is not necessary except for families invited for additional testing.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include all individuals with a combination of medical problems including muscle and bone disease and their family members. Because historically VCP related muscle disease has been erroneously diagnosed with the following diagnoses, therefore if these patients also have a personal or family history of bone disease they will be considered eligible for the study:

Muscle disorders considered include:

* Limb Girdle Muscular Dystrophy
* Myopathy
* Inclusion body myopathy
* FSH (Facioscapular muscular dystrophy) without the mutation
* Scapuloperoneal muscular dystrophy
* Amyotrophic Lateral Sclerosis
* Non specific muscular dystrophy

AND

* Bone disorders including:

  * Paget disease of bone
  * Fibrous dysplasia
  * Diaphyseal medullary stenosis with malignant fibrous histiocytoma (DMS-MFH)
  * Non-specific bone disease

Eligible participants must also be:

* Subjects must to 18 years or older
* Subjects must to able to give consent
* Adult family members or spouses over the age of 18 of the affected individuals

Exclusion Criteria:

* Under the age of 18.

Individuals who report a different unrelated diagnosis will be excluded from the study. Testing to confirm different diagnoses will not be performed, instead patient will be questioned for this information and records will be obtained for confirmation of appropriate testing.

Those who are unable to provide consent for themselves will be excluded from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with a personal or family history of VCP associated disease.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-11-15 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kimonis, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

REFERENCES:
- [Background] Kimonis VE, Fulchiero E, Vesa J, Watts G. VCP disease associated with myopathy, Paget disease of bone and frontotemporal dementia: review of a unique disorder. Biochim Biophys Acta. 2008 Dec;1782(12):744-8. doi: 10.1016/j.bbadis.2008.09.003. Epub 2008 Sep 18. PMID 18845250
- [Background] Llewellyn KJ, Walker N, Nguyen C, Tan B, BenMohamed L, Kimonis VE, Nalbandian A. A Fine Balance of Dietary Lipids Improves Pathology of a Murine Model of VCP-Associated Multisystem Proteinopathy. PLoS One. 2015 Jul 2;10(7):e0131995. doi: 10.1371/journal.pone.0131995. eCollection 2015. PMID 26134519
- [Result] Tresse E, Salomons FA, Vesa J, Bott LC, Kimonis V, Yao TP, Dantuma NP, Taylor JP. VCP/p97 is essential for maturation of ubiquitin-containing autophagosomes and this function is impaired by mutations that cause IBMPFD. Autophagy. 2010 Feb;6(2):217-27. doi: 10.4161/auto.6.2.11014. Epub 2010 Feb 22. PMID 20104022
- [Result] Hubbers CU, Clemen CS, Kesper K, Boddrich A, Hofmann A, Kamarainen O, Tolksdorf K, Stumpf M, Reichelt J, Roth U, Krause S, Watts G, Kimonis V, Wattjes MP, Reimann J, Thal DR, Biermann K, Evert BO, Lochmuller H, Wanker EE, Schoser BG, Noegel AA, Schroder R. Pathological consequences of VCP mutations on human striated muscle. Brain. 2007 Feb;130(Pt 2):381-93. doi: 10.1093/brain/awl238. Epub 2006 Sep 19. PMID 16984901
- [Result] Vesa J, Su H, Watts GD, Krause S, Walter MC, Martin B, Smith C, Wallace DC, Kimonis VE. Valosin containing protein associated inclusion body myopathy: abnormal vacuolization, autophagy and cell fusion in myoblasts. Neuromuscul Disord. 2009 Nov;19(11):766-72. doi: 10.1016/j.nmd.2009.08.003. Epub 2009 Oct 13. PMID 19828315
- [Result] Weihl CC, Pestronk A, Kimonis VE. Valosin-containing protein disease: inclusion body myopathy with Paget's disease of the bone and fronto-temporal dementia. Neuromuscul Disord. 2009 May;19(5):308-15. doi: 10.1016/j.nmd.2009.01.009. Epub 2009 Apr 19. PMID 19380227
- [Result] Kimonis VE, Mehta SG, Fulchiero EC, Thomasova D, Pasquali M, Boycott K, Neilan EG, Kartashov A, Forman MS, Tucker S, Kimonis K, Mumm S, Whyte MP, Smith CD, Watts GD. Clinical studies in familial VCP myopathy associated with Paget disease of bone and frontotemporal dementia. Am J Med Genet A. 2008 Mar 15;146A(6):745-57. doi: 10.1002/ajmg.a.31862. PMID 18260132
- [Result] Watts GD, Thomasova D, Ramdeen SK, Fulchiero EC, Mehta SG, Drachman DA, Weihl CC, Jamrozik Z, Kwiecinski H, Kaminska A, Kimonis VE. Novel VCP mutations in inclusion body myopathy associated with Paget disease of bone and frontotemporal dementia. Clin Genet. 2007 Nov;72(5):420-6. doi: 10.1111/j.1399-0004.2007.00887.x. PMID 17935506
- [Result] Mehta SG, Watts GD, Adamson JL, Hutton M, Umberger G, Xiong S, Ramdeen S, Lovell MA, Kimonis VE, Smith CD. APOE is a potential modifier gene in an autosomal dominant form of frontotemporal dementia (IBMPFD). Genet Med. 2007 Jan;9(1):9-13. doi: 10.1097/gim.0b013e31802d830d. PMID 17224685
- [Result] Forman MS, Mackenzie IR, Cairns NJ, Swanson E, Boyer PJ, Drachman DA, Jhaveri BS, Karlawish JH, Pestronk A, Smith TW, Tu PH, Watts GD, Markesbery WR, Smith CD, Kimonis VE. Novel ubiquitin neuropathology in frontotemporal dementia with valosin-containing protein gene mutations. J Neuropathol Exp Neurol. 2006 Jun;65(6):571-81. doi: 10.1097/00005072-200606000-00005. PMID 16783167
- [Result] Mehta SG, Watts GD, McGillivray B, Mumm S, Hamilton SJ, Ramdeen S, Novack D, Briggs C, Whyte MP, Kimonis VE. Manifestations in a family with autosomal dominant bone fragility and limb-girdle myopathy. Am J Med Genet A. 2006 Feb 15;140(4):322-30. doi: 10.1002/ajmg.a.31008. PMID 16419137
- [Result] Kimonis VE, Watts GD. Autosomal dominant inclusion body myopathy, Paget disease of bone, and frontotemporal dementia. Alzheimer Dis Assoc Disord. 2005 Oct-Dec;19 Suppl 1:S44-7. doi: 10.1097/01.wad.0000183081.76820.5a. PMID 16317258
- [Result] Lucas GJ, Mehta SG, Hocking LJ, Stewart TL, Cundy T, Nicholson GC, Walsh JP, Fraser WD, Watts GD, Ralston SH, Kimonis VE. Evaluation of the role of Valosin-containing protein in the pathogenesis of familial and sporadic Paget's disease of bone. Bone. 2006 Feb;38(2):280-5. doi: 10.1016/j.bone.2005.07.014. Epub 2005 Sep 30. PMID 16199218
- [Result] Watts GD, Wymer J, Kovach MJ, Mehta SG, Mumm S, Darvish D, Pestronk A, Whyte MP, Kimonis VE. Inclusion body myopathy associated with Paget disease of bone and frontotemporal dementia is caused by mutant valosin-containing protein. Nat Genet. 2004 Apr;36(4):377-81. doi: 10.1038/ng1332. Epub 2004 Mar 21. PMID 15034582
- [Result] Watts GD, Thorne M, Kovach MJ, Pestronk A, Kimonis VE. Clinical and genetic heterogeneity in chromosome 9p associated hereditary inclusion body myopathy: exclusion of GNE and three other candidate genes. Neuromuscul Disord. 2003 Sep;13(7-8):559-67. doi: 10.1016/s0960-8966(03)00070-1. PMID 12921793
- [Result] Kimonis V. Inclusion Body Myopathy with Paget Disease of Bone and/or Frontotemporal Dementia. 2007 May 25 [updated 2019 Sep 12]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1476/ PMID 20301649
- [Result] Plewa J, Surampalli A, Wencel M, Milad M, Donkervoort S, Caiozzo VJ, Goyal N, Mozaffar T, Kimonis V. A cross-sectional analysis of clinical evaluation in 35 individuals with mutations of the valosin-containing protein gene. Neuromuscul Disord. 2018 Sep;28(9):778-786. doi: 10.1016/j.nmd.2018.06.007. Epub 2018 Jun 27. PMID 30097247
- [Result] Al-Tahan S, Al-Obeidi E, Yoshioka H, Lakatos A, Weiss L, Grafe M, Palmio J, Wicklund M, Harati Y, Omizo M, Udd B, Kimonis V. Novel valosin-containing protein mutations associated with multisystem proteinopathy. Neuromuscul Disord. 2018 Jun;28(6):491-501. doi: 10.1016/j.nmd.2018.04.007. Epub 2018 Apr 17. PMID 29754758
- [Result] Al-Obeidi E, Al-Tahan S, Surampalli A, Goyal N, Wang AK, Hermann A, Omizo M, Smith C, Mozaffar T, Kimonis V. Genotype-phenotype study in patients with valosin-containing protein mutations associated with multisystem proteinopathy. Clin Genet. 2018 Jan;93(1):119-125. doi: 10.1111/cge.13095. PMID 28692196
- [Result] Llewellyn KJ, Nalbandian A, Weiss LN, Chang I, Yu H, Khatib B, Tan B, Scarfone V, Kimonis VE. Myogenic differentiation of VCP disease-induced pluripotent stem cells: A novel platform for drug discovery. PLoS One. 2017 Jun 2;12(6):e0176919. doi: 10.1371/journal.pone.0176919. eCollection 2017. PMID 28575052
- [Result] Evangelista T, Weihl CC, Kimonis V, Lochmuller H; VCP related diseases Consortium. 215th ENMC International Workshop VCP-related multi-system proteinopathy (IBMPFD) 13-15 November 2015, Heemskerk, The Netherlands. Neuromuscul Disord. 2016 Aug;26(8):535-47. doi: 10.1016/j.nmd.2016.05.017. Epub 2016 May 30. No abstract available. PMID 27312024
- [Result] Rodriguez-Ortiz CJ, Flores JC, Valenzuela JA, Rodriguez GJ, Zumkehr J, Tran DN, Kimonis VE, Kitazawa M. The Myoblast C2C12 Transfected with Mutant Valosin-Containing Protein Exhibits Delayed Stress Granule Resolution on Oxidative Stress. Am J Pathol. 2016 Jun;186(6):1623-34. doi: 10.1016/j.ajpath.2016.02.007. Epub 2016 Apr 20. PMID 27106764
- [Result] Nalbandian A, Llewellyn KJ, Gomez A, Walker N, Su H, Dunnigan A, Chwa M, Vesa J, Kenney MC, Kimonis VE. In vitro studies in VCP-associated multisystem proteinopathy suggest altered mitochondrial bioenergetics. Mitochondrion. 2015 May;22:1-8. doi: 10.1016/j.mito.2015.02.004. Epub 2015 Feb 25. PMID 25724235
- [Result] Surampalli A, Khare M, Kubrussi G, Wencel M, Tanaja J, Donkervoort S, Osann K, Simon M, Wallace D, Smith C, M McInerney-Leo A, Kimonis V. Psychological Impact of Predictive Genetic Testing in VCP Inclusion Body Myopathy, Paget Disease of Bone and Frontotemporal Dementia. J Genet Couns. 2015 Oct;24(5):842-50. doi: 10.1007/s10897-015-9819-7. Epub 2015 Feb 26. PMID 25716352
- [Result] Surampalli A, Gold BT, Smith C, Castellani RJ, Khare M, Yu H, Nguyen C, Lan M, Wencel M, Wigal S, Caiozzo V, Kimonis V. A case report comparing clinical, imaging and neuropsychological assessment findings in twins discordant for the VCP p.R155C mutation. Neuromuscul Disord. 2015 Feb;25(2):177-83. doi: 10.1016/j.nmd.2014.10.003. Epub 2014 Oct 22. PMID 25582679
- [Result] Shamirian S, Nalbandian A, Khare M, Castellani R, Kim R, Kimonis VE. Early-onset Alzheimers and cortical vision impairment in a woman with valosin-containing protein disease associated with 2 APOE epsilon4/APOE epsilon4 genotype. Alzheimer Dis Assoc Disord. 2015 Jan-Mar;29(1):90-3. doi: 10.1097/WAD.0b013e318298e54f. PMID 23715207
- [Result] Kim HJ, Kim NC, Wang YD, Scarborough EA, Moore J, Diaz Z, MacLea KS, Freibaum B, Li S, Molliex A, Kanagaraj AP, Carter R, Boylan KB, Wojtas AM, Rademakers R, Pinkus JL, Greenberg SA, Trojanowski JQ, Traynor BJ, Smith BN, Topp S, Gkazi AS, Miller J, Shaw CE, Kottlors M, Kirschner J, Pestronk A, Li YR, Ford AF, Gitler AD, Benatar M, King OD, Kimonis VE, Ross ED, Weihl CC, Shorter J, Taylor JP. Mutations in prion-like domains in hnRNPA2B1 and hnRNPA1 cause multisystem proteinopathy and ALS. Nature. 2013 Mar 28;495(7442):467-73. doi: 10.1038/nature11922. Epub 2013 Mar 3. PMID 23455423
- [Result] Mehta SG, Khare M, Ramani R, Watts GD, Simon M, Osann KE, Donkervoort S, Dec E, Nalbandian A, Platt J, Pasquali M, Wang A, Mozaffar T, Smith CD, Kimonis VE. Genotype-phenotype studies of VCP-associated inclusion body myopathy with Paget disease of bone and/or frontotemporal dementia. Clin Genet. 2013 May;83(5):422-31. doi: 10.1111/cge.12000. Epub 2012 Oct 4. PMID 22909335
- [Result] Nalbandian A, Ghimbovschi S, Radom-Aizik S, Dec E, Vesa J, Martin B, Knoblach S, Smith C, Hoffman E, Kimonis VE. Global gene profiling of VCP-associated inclusion body myopathy. Clin Transl Sci. 2012 Jun;5(3):226-34. doi: 10.1111/j.1752-8062.2012.00407.x. Epub 2012 Apr 4. PMID 22686199
- [Result] Nalbandian A, Donkervoort S, Dec E, Badadani M, Katheria V, Rana P, Nguyen C, Mukherjee J, Caiozzo V, Martin B, Watts GD, Vesa J, Smith C, Kimonis VE. The multiple faces of valosin-containing protein-associated diseases: inclusion body myopathy with Paget's disease of bone, frontotemporal dementia, and amyotrophic lateral sclerosis. J Mol Neurosci. 2011 Nov;45(3):522-31. doi: 10.1007/s12031-011-9627-y. Epub 2011 Sep 3. PMID 21892620
- [Result] Chan N, Le C, Shieh P, Mozaffar T, Khare M, Bronstein J, Kimonis V. Valosin-containing protein mutation and Parkinson's disease. Parkinsonism Relat Disord. 2012 Jan;18(1):107-9. doi: 10.1016/j.parkreldis.2011.07.006. Epub 2011 Aug 3. No abstract available. PMID 21816654
- [Result] Farpour F, Tehranzadeh J, Donkervoort S, Smith C, Martin B, Vanjara P, Osann K, Kimonis VE. Radiological features of Paget disease of bone associated with VCP myopathy. Skeletal Radiol. 2012 Mar;41(3):329-37. doi: 10.1007/s00256-011-1193-4. Epub 2011 Jun 4. PMID 21643886
- [Result] Fanganiello RD, Kimonis VE, Corte CC, Nitrini R, Passos-Bueno MR. A Brazilian family with hereditary inclusion body myopathy associated with Paget disease of bone and frontotemporal dementia. Braz J Med Biol Res. 2011 Apr;44(4):374-80. doi: 10.1590/s0100-879x2011007500028. Epub 2011 Mar 11. PMID 21412659
- [Derived] Shmara A, Perez-Rosendahl M, Murphy K, Kwon A, Smith C, Kimonis V. A clinicopathologic study of malignancy in VCP-associated multisystem proteinopathy. Orphanet J Rare Dis. 2022 Jul 15;17(1):272. doi: 10.1186/s13023-022-02403-9. PMID 35841038
- See also: Bibliography — https://www.ncbi.nlm.nih.gov/pubmed/?term=kimonis+v